CLINICAL TRIAL: NCT04582513
Title: Impact of an Anesthesia Care Handover-Checklist on Adverse Perioperative Outcome (AnCHor - Checklist) Pilot Trial
Brief Title: Impact of an Anesthesia Care Handover-Checklist on Adverse Perioperative Outcome
Acronym: AnCHor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Jan Larmann, Attending Anaesthesiologist, University Hospital Heidelberg
Other Study IDs: AnCHor
Record Dates: First submitted 2020-09-26; First posted 2020-10-09 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Major Surgery
Keywords: handover; anaesthesia; checklist; perioperative complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-checklist implementation group: Patients undergoing major elective surgery where intraoperative handover occurs. This handover is performed according to current hospital standard without a standardized checklist.
- Post-checklist implementation group: Patients undergoing major elective surgery where intraoperative handover occurs. This handover is performed after implementation of the AnCHor-CHecklist, a standardized checklist based on the SBAR concept.
  Interventions: Other: AnCHor-Checklist implementation

INTERVENTIONS:
Other: AnCHor-Checklist implementation — a standardized checklist using the SBAR concept according to the recommendations of the DGAI
  Groups: Post-checklist implementation group

SUMMARY:
The aim of the study is to collect information on feasibility and effect size of a confirmatory, prospective study with the question: Does a standardized checklist during intraoperative handover of anaesthesia care reduce the rate of postoperative complications?

DETAILED DESCRIPTION:
During clinical routine, intraoperative handover of anaesthesia care occurs frequently. This handover between two anaesthesiologists requires the transmission of all relevant information concerning the patient and the ongoing procedure. Studies regarding the influence of such handovers on patient outcome are inconclusive and mostly of retrospective nature. Some studies report a negative effect of handovers on patients mortality and outcome, however studies exist reporting no effect. A positive effect of intraoperative handovers as a result of a "second man" effect ist also possible. To increase handover quality, the German Society of Anaesthesiology and Intensive Care Medicine (DGAI) recommends the application of the situation, background, assessment and recommendation (SBAR) concept. Information are arranged in those four groups with the goal of structuring the handover and incorporating all relevant information. Studies show increased accuracy of transferred information and improved comprehensibility when using the SBAR concept. Whether an intraoperative handover according to the SBAR concept reduces the rate of postoperative complications is not yet investigated. Due to lack of information regarding feasibility and effect size, the investigators plan a prospective pilot study to answer these questions. Initially, patients undergoing major surgery are recruited where handover is performed without a standardized handover. After the implementation of a checklist using the SBAR concept, this checklist will be used during intraoperative handover in recruited patients where a handover occurs. The primary endpoint is a combined endpoint consisting of all-cause mortality, readmission to any hospital, or major postoperative complications. Additionally, implementation rate and efficacy of the checklist will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Major surgeries with a duration of at least 2 h (requirement of postoperative admission to hospital for at least 1 night)
* American Society of Anesthesiologists (ASA) Classification 3-4
* Informed consent

Exclusion Criteria:

* Patients incapable of consent
* Previous surgery within the same surgical subgroup within the last 6 months
* Pregnancy, breastfeeding
* Patients participating in another interventional trial within the last 3 months with possible interference to the outcome of this study
* Persons with any kind of dependency on the investigator or employed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective major non cardiac surgery, admitted to University Hospital Heidelberg
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Composite of mortality, hospital readmission and major postoperative complications | within 30 days of index surgery
  Number of patients that die and/or are readmitted to any hospital and/or experience any of the following: prolonged postoperative ventilation >48 hours, major disruption of surgical wound, bleeding, pneumonia, atrial fibrillation, moderate or severe acute kidney injury, new onset of hemodialysis, cardiac arrest, myocardial infarction, sepsis, stroke, pulmonary embolism, deep venous thrombosis, shock, unplanned return to operating room

SECONDARY OUTCOMES:
Implementation of checklist | on day of index surgery
  Rate of correctly filed checklists
Determination of recruitment rate | within 30 days of index surgery
  Rate of recruited patients in all recruitable patients
Prolonged postoperative Ventilation >48 hours | within 48 hours after index surgery
  Number of patients with prolonged postoperative ventilation defined as ≥ 48h need of invasive mechanical ventilation via endotracheal tube or need for tracheostomy due to prolonged weaning
Major disruption of surgical wound | within 30 days of index surgery
  Number of patients with major disruption of surgical wound defined as the need for re-operation (wound dehiscence, burst abdomen)
Bleeding | within the initial surgical procedure and within 30 days after index surgery
  Number of patients with bleeding complications defined as major bleeding with transfusion requirement and/ or the need for re-operation (hematothorax, relaparotomy, and removal of hematoma)
Insufficiency of anastomoses | within 30 days of index surgery
  Number of patients with insufficiency of anastomoses defined by International Study Group of Rectal Cancer (ISREC)-definition
Intra-abdominal abcess | within 30 days of index surgery
  Number of patients with intra-abdominal abscess defined by imaging
Pneumonia | within 30 days of index surgery
  Number of patients with pneumonia defined as occurence of pneumonia verified by X-ray
Atrial fibrillation | within 30 days of index surgery
  Number of patients with atrial fibrillation defined as new onset of atrial fibrillation without any known episode prior to index surgery
Occurrence of moderate or severe acute kidney injury | within 30 days after index surgery
  Number of patients with moderate acute kidney injury (AKI) defined as Kidney Disease: Improving Global Outcomes (KDIGO) stage 2 (≥ 2-fold increase in serum-creatinine from baseline and/or urine output < 0.5 ml/kg/h for ≥ 12 h) or severe AKI is defined as KDIGO stage 3 (≥ 3-fold serum creatinine increase from baseline and/or urine output ≤ 0.3 ml/kg/h for ≥ 24 h)
New onset of hemodialysis | within 30 days after index surgery
  Number of patients with new onset of need for renal replacement therapy
Cardiac arrest | within 30 days of index surgery
  Number of patients with cardiac arrest defined as the need for cardiopulmonary resuscitation
Myocardial infarction | during index surgery and within 30 days after index surgery
  Number of patients with myocardial infarction defined by by ST elevation in the ECG and/or troponin elevation in patients with acute chest pain
Sepsis | within 30 days of index surgery
  Number of patients with sepsis defined according to Sepsis3 guidelines
Stroke | within 30 days of index surgery
  Number of patients with stroke defined by verification in a CT scan
Pulmonary embolism and deep venous thromboembolism | within 30 days of index surgery
  Number of patients with pulmonary embolism and deep venous thromboembolism defined by verification in a CT scan
Shock | during the initial surgical procedure and within 30 days after index surgery
  Number of patients with shock defined based on the corresponding International Statistical Classification of Diseases and Related Health Problems (ICD-10) codes (R57.1, R57.8, R57.9)
unplanned return to operating room | within 30 days of index surgery
  Number of patients with unplanned return to operating room within time frame
Need for intervention | within 30 days of index surgery
  Number of patients with interventions defined as endoscopy, Insertion of drains or stents
Hospital length of stay | within 30 days of index surgery
  Documented in patient charts
ICU admission | within 30 days of index surgery
  Number of patients with ICU admission
ICU length of stay | within 30 days of index surgery
  Documented in patient charts
total morbidity | within 30 days of index surgery
  defined by Comprehensive Complication Index (CCI)
All-cause mortality | within 30 days of index surgery
  Number of patients died within 30 days of index surgery
Readmission to any hospital | within 30 days of index surgery
  Number of patients with any readmission to an acute care hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jan Larmann, MD PhD, Principal Investigator — Departement of Anaesthesiology, Heidelberg University Hospital
Locations (1):
- Department of Anaesthesiology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones PM, Cherry RA, Allen BN, Jenkyn KMB, Shariff SZ, Flier S, Vogt KN, Wijeysundera DN. Association Between Handover of Anesthesia Care and Adverse Postoperative Outcomes Among Patients Undergoing Major Surgery. JAMA. 2018 Jan 9;319(2):143-153. doi: 10.1001/jama.2017.20040. PMID 29318277
- [Background] Hudson CC, McDonald B, Hudson JK, Tran D, Boodhwani M. Impact of anesthetic handover on mortality and morbidity in cardiac surgery: a cohort study. J Cardiothorac Vasc Anesth. 2015 Feb;29(1):11-6. doi: 10.1053/j.jvca.2014.05.018. Epub 2014 Nov 24. PMID 25440620
- [Background] Saager L, Hesler BD, You J, Turan A, Mascha EJ, Sessler DI, Kurz A. Intraoperative transitions of anesthesia care and postoperative adverse outcomes. Anesthesiology. 2014 Oct;121(4):695-706. doi: 10.1097/ALN.0000000000000401. PMID 25102312
- [Background] Terekhov MA, Ehrenfeld JM, Dutton RP, Guillamondegui OD, Martin BJ, Wanderer JP. Intraoperative Care Transitions Are Not Associated with Postoperative Adverse Outcomes. Anesthesiology. 2016 Oct;125(4):690-9. doi: 10.1097/ALN.0000000000001246. PMID 27466034
- [Background] McCrory MC, Aboumatar H, Custer JW, Yang CP, Hunt EA. "ABC-SBAR" training improves simulated critical patient hand-off by pediatric interns. Pediatr Emerg Care. 2012 Jun;28(6):538-43. doi: 10.1097/PEC.0b013e3182587f6e. PMID 22653454
- [Background] Randmaa M, Martensson G, Leo Swenne C, Engstrom M. SBAR improves communication and safety climate and decreases incident reports due to communication errors in an anaesthetic clinic: a prospective intervention study. BMJ Open. 2014 Jan 21;4(1):e004268. doi: 10.1136/bmjopen-2013-004268. PMID 24448849
- [Background] Agarwala AV, Firth PG, Albrecht MA, Warren L, Musch G. An electronic checklist improves transfer and retention of critical information at intraoperative handoff of care. Anesth Analg. 2015 Jan;120(1):96-104. doi: 10.1213/ANE.0000000000000506. PMID 25625256
- [Background] Marshall S, Harrison J, Flanagan B. The teaching of a structured tool improves the clarity and content of interprofessional clinical communication. Qual Saf Health Care. 2009 Apr;18(2):137-40. doi: 10.1136/qshc.2007.025247. PMID 19342529